CLINICAL TRIAL: NCT05437146
Title: The Effect of Therapeutic Play Applied With Puppet During Blood Collection in Children on Pain and Fear
Brief Title: The Effect of Therapeutic Play Applied With Puppet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/449
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Bloodletting

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puppet (Experimental): pain and fear
  Interventions: Behavioral: puppet
- control (No Intervention): not pain and fear

INTERVENTIONS:
Behavioral: puppet — pain and fear during blood collection
  Arms: Puppet

SUMMARY:
The aim of this study is to determine the effect of therapeutic play applied with a hand puppet during blood collection on pain and fear in children. The project is a randomized controlled trial. The study includes children aged 3-6 years who came to the pediatric blood collection unit of Binali Yıldırım University Mengücek Gazi Training and Research Hospital between 01/07/2022 and 01/01/2023. The research sample; children who apply to the unit on the specified dates and meet the research criteria and volunteer to participate in the research. "Survey Form", "Wong-Baker Evaluation of Facial Expressions Scale" and "Child Fear Scale" will be used in data collection.

DETAILED DESCRIPTION:
Type of Study: The study is a randomized controlled trial. Population and Sample of the Research: The population of the research includes children aged 3-6 years who came to the pediatric blood collection unit of Binali Yıldırım University Mengücek Gazi Training and Research Hospital between 01/07/2022-01/01/2023.

The research sample; "Children who apply to the blood collection unit on the specified dates and meet the research criteria and volunteer to participate in the research". In this study, "prior power analysis" was conducted to determine sample adequacy. In the Priori power analysis, "Cohen's method of reference to standard effect sizes" was chosen. In this case, in our study, the effect of the therapeutic game applied with a hand puppet during blood collection on pain and fear in children will be compared. It has been determined that 80% power can be reached. It was decided to collect data from a total of 100 individuals by including 10% backup sample in this number in case of data loss. Data collection will not be carried out simultaneously in the puppet and control groups, in case the children in the clinic are affected by the puppet toys. In order to ensure randomization, the children who met the criteria will be included in the control group in the first week, and the children who come in the second week will be taken into the puppet group, and this cycle will be continued until the end of the study, and randomization will be ensured.

Data Collection Tools to be Used in the Study: "Survey Form, Wong-Baker Facial Expression Evaluation Scale and Child Fear Scale" will be used to collect research data. As an intervention tool in the research, a hand puppet designed together with the researcher and child development specialist will be used.

Questionnaire Form: In the questionnaire form created by the researchers by scanning the literature; There are questions addressing the introductory characteristics of the research group.

Intervention Tools to be Used in the Research Hand puppet: A hand puppet designed together with the researcher and child development specialist will be used as an intervention tool in the research. In this context, the researcher received play therapy training. While the puppet is being designed, it will be ensured that it is integrated in the hospital environment and it will be ensured that the child is not alienated to the environment he/she comes from. The researcher, who received play therapy training in hand puppet practice, plans to reduce the children's fears and reduce the level of pain before the intervention. While designing the hand puppet, care will be taken to ensure that the materials to be used are antiallergenic and made of fabric that can be easily sterilized after each child the application is made.

Data Collection The researcher will stay in the pediatric blood collection unit for 1 day in order to examine the ergonomic structure of the pediatric blood collection unit before collecting the data of the puppet group and control group children. Parents were informed about the research (the purpose of the research, why the research was conducted, the use of a puppet toy to relieve the child's pain and fear, etc.), after giving verbal consent from the children and written consent from the parents. Afterwards, the data of the research will be obtained by face-to-face interview method with the children who accepted to participate in the research.

Control Group: Questionnaires and scales will be filled in the control group 5 minutes before the blood draw is done by the researcher. Only routine applications will be made. 5 minutes after the procedure, the scales will be filled again. Filling out the forms will take 5-10 minutes on average.

Puppet Group: Questionnaires and scales will be filled in 5 minutes before the blood draw is done by the researcher. It will be played with the puppet during the process. 5 minutes after the procedure, the scales will be filled again. Filling out the forms will take 5-10 minutes on average.

Evaluation of Data The processing and statistical analysis of the collected data will be done with the analysis software called SPSS (Statistical Package for the Social Sciences) for Windows 20.0.

Ethical Principles of Research In order to carry out the research, official permission from the relevant institution will be obtained from the Ethics Committee with ethical approval. Children who meet the criteria of the research group will be informed about the purpose of the study, their questions will be answered, and their verbal and written consent will be obtained. Parents and children will be informed that the data collected during the research will be processed anonymously, confidentially, and will not be used outside of the study in question, and that they can leave the study whenever they wish. Since the research is based on the use of data obtained from humans, and therefore, due to the necessity of observing personal rights, the relevant ethical principles "Informed Consent", "Volunteerism" and "Protection of Confidentiality" will be followed. After the blood collection process is completed, the children in the control group will be played with a puppet and the "Principle of Equality" will be tried to be fulfilled.

ELIGIBILITY:
Inclusion Criteria:

* be between 3-6 years old
* Not having a disability related to developmental areas
* Not taking analgesics within 24 hours before application
* Being with the mother or father of the child during the procedure

Exclusion Criteria:

* Not between 3-6 years old
* Having a disability related to developmental areas
* Taking analgesics within 24 hours before admission
* Not being with the mother or father of the child during the procedure

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-06-19 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Evaluation Scale (WB-FAI) | 9 MONTHS
  The scale was developed in 1981 and was revised in 1983. The scale is used to define pain in the 3-18 age group. The scale indicates that the severity of pain increases from zero to five as you go from left to right. Facial expressions are included under the numbers to describe the severity of pain. It consists of 6 faces in total. While the first smiling facial expression expresses the pain-free state, the crying facial expression at the end indicates the most severe pain intensity. While applying the scale, the child is told to choose the facial expression that best describes his feelings at the moment. Six facial expressions are scored between 0-5 points from left to right (0 points = very happy/no pain, 5 points = indicates the most severe pain). As the score obtained from the scale increases, the pain tolerance decreases, and as the score decreases, the tolerance increases.
Child Fear Scale (CFS): | 9 MONTHS
  The scale was developed in 2011. The Child Fear Scale is used to determine the level of fear in children undergoing painful medical procedures. The Child Fear Scale is a scale from 0-4 showing five faces ranging from a neutral expression (0 = no worry) to the feared face (4 = serious anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Study Director — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED